CLINICAL TRIAL: NCT05750277
Title: The Feasibility of Early Time-Restricted Eating in a Student Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nottingham Trent University (Other)
Responsible Party: Principal Investigator, William Mode, Principal Investigator, Nottingham Trent University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NottinghamTU1
Record Dates: First submitted 2023-02-02; First posted 2023-03-01 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Time Restricted Feeding; Intermittent Fasting
Keywords: Students; Metabolism; Appetite
MeSH Terms: conditions — Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Time-Restricted Eating (Experimental): This group will self-select their eating window as long as it is between 8am-6pm, and will aim to fast within this window as many occasions as possible between Monday-Friday for 4 weeks.
  Interventions: Other: Evening Time-Restricted Eating
- Control (No Intervention): This group will maintain their habitual lifestyle for 4 weeks.

INTERVENTIONS:
Other: Evening Time-Restricted Eating — Eating between 8am-6pm.
  Arms: Early Time-Restricted Eating

SUMMARY:
This study proposes to investigate the effect of a self-selected early time-restricted eating window in University students.

DETAILED DESCRIPTION:
There were over 2.3 million students registered at Higher Education institutes in the UK. Early adulthood is a critical time for establishing self-care habits which will ultimately influence health outcomes later in adulthood and studies suggest that the overall health of students is poor relative to that of their age-matched peers not in education. Therefore, the investigators would like to assess the feasibility of adopting a novel, nutritional intervention in this important, understudied population.

Previous research has shown Early Time-Restricted Eating can reduce daily energy consumed and improve markers of health over time, in a range of populations. Therefore, the investigators are investigating how often participants can eat within an early 8 hour eating window, starting no earlier than 8am (finishing calorie intake by 4pm), or no later than 10am (finishing calorie intake by 6pm). The investigators will be measuring how often the participants can adhere to this eating window between Monday to Friday, with the study lasting 4 weeks in total. This is a feasibility study, so this study will investigate whether this intervention is achievable and what social barriers may exist which reduce adherence to this eating window. Participants will visit the laboratory on 3 occasions (at the start, halfway point, and at the end of the intervention) to measure any changes in health markers across the intervention. The lab visits will involve providing a finger-tip blood sample, and measuring body mass, blood pressure, and waist-to-hip circumference. Outside of the laboratory, participants are required to record their eating window on a mobile app and an investigator-created trial sheet. Further measures outside of the laboratory will include a weekly questionnaire and motivational correspondence via mobile text message.

ELIGIBILITY:
Inclusion Criteria:

* Registered student

Exclusion Criteria:

* Not taking any medication which is known to affect appetite

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-04-19 (Actual); Primary Completion 2023-05-18 (Estimated); Study Completion 2023-05-19 (Estimated)

PRIMARY OUTCOMES:
Successful bouts of Early Time-Restricted Eating | 4 weeks
  Successful Early Time-Restricted Eating occasions will be recorded by the participant on a mobile device and an investigator-created trial sheet.

SECONDARY OUTCOMES:
Glucose | 4 weeks
  How their glucose concentrations change over the trial
Insulin | 4 weeks
  How their Insulin concentrations change over the trial
HbA1C | 4 weeks
  How their HbA1CA concentrations change over the trial
Body mass | 4 weeks
  How their body mass changes over the trial
Blood pressure | 4 weeks
  How blood pressure (systolic and diastolic) changes over the trial
Body fat percentage | 4 weeks
  How their body fat percentage changes over the trial
Waist to hip ratio | 4 weeks
  How their waist to hip ratio changes over the trial
Appetite | 4 weeks
  Investigators will record appetite sensations, such as; hunger, fullness, prospective food consumption, desire to eat and nausea. Investigators will record these validated sensations to observe any changes across the trial. A visual analogue scale (100mm) will be digitised and sent to the participant by mobile text to record changes in the aforementioned appetitte sensations.

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham Trent University, Nottingham, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No